CLINICAL TRIAL: NCT03680638
Title: The Effect of Antioxidants on Skin Blood Flow During Local Heating
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Associate Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-0268
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Vasodilation
Keywords: Racial Differences; Oxidative Stress; Obesity; Local Heating
MeSH Terms: conditions — Cardiovascular Diseases; Aneurysm; Obesity | interventions — Ringer's Lactate; tempol; acetovanillone; Allopurinol

STUDY DESIGN:
Intervention Model Description: Each subject has one control site and three experimental sites concurrently tested within the same study using intradermal microdialysis on the dorsal forearm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control (Lactated Ringer's) (Sham Comparator): This site will only be infused with Lactated Ringer's during the local heating stimulus. After the local heating stimulus, this site will be infused with L-NAME (Nω-nitro-L-arginine methylester; 20mM) to inhibit nitric oxide synthase and with SNP (sodium nitroprusside; 28mM) to elicit vasodilation. This will help establish nitric oxide contribution to vasodilation and establish maximal vasodilation for data normalization, respectively.
  Interventions: Other: Control (Lactated Ringer's)
- Tempol (Experimental): This site will only be infused with tempol (4-hydroxy-2,2,6,6-tetramethylpiperidine-1-oxyl; 10µM) during the local heating stimulus. After the local heating stimulus, this site will be infused with L-NAME (Nω-nitro-L-arginine methylester; 20mM) to inhibit nitric oxide synthase and with SNP (sodium nitroprusside; 28mM) to elicit vasodilation. This will help establish nitric oxide contribution to vasodilation and establish maximal vasodilation for data normalization, respectively.
  Interventions: Drug: Tempol
- Apocynin (Experimental): This site will only be infused with apocynin (1-(4-Hydroxy-3-methoxyphenyl)ethanone; 100µM) during the local heating stimulus. After the local heating stimulus, this site will be infused with L-NAME (Nω-nitro-L-arginine methylester; 20mM) to inhibit nitric oxide synthase and with SNP (sodium nitroprusside; 28mM) to elicit vasodilation. This will help establish nitric oxide contribution to vasodilation and establish maximal vasodilation for data normalization, respectively.
  Interventions: Drug: Apocynin
- Allopurinol (Experimental): This site will only be infused with tempol (1H-pyrazolo[3,4-d]pyrimidin-4(2H)-one; 10µM) during the local heating stimulus. After the local heating stimulus, this site will be infused with L-NAME (Nω-nitro-L-arginine methylester; 20mM) to inhibit nitric oxide synthase and with SNP (sodium nitroprusside; 28mM) to elicit vasodilation. This will help establish nitric oxide contribution to vasodilation and establish maximal vasodilation for data normalization, respectively.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Other: Control (Lactated Ringer's) — This intervention is meant to serve as a control by which the experimental sites are compared to, to assess effectiveness.
  Arms: Control (Lactated Ringer's)
Drug: Tempol — This intervention is meant to assess the impact of superoxide on vasodilator responses by scavenging available superoxide.
  Arms: Tempol
Drug: Apocynin — This intervention is meant to assess the impact of NADPH oxidase-derived superoxide on vasodilator responses by inhibiting the enzyme NADPH oxidase.
  Arms: Apocynin
Drug: Allopurinol — This intervention is meant to assess the impact of xanthine oxidase-derived superoxide on vasodilator responses by inhibiting the enzyme xanthine oxidase.
  Arms: Allopurinol

SUMMARY:
The goal of this study is to examine possible mechanisms of impaired vasodilaton in obese and Black/African American men and women as possible links to the elevated prevalence of cardiovascular dysfunction and disease. The main targets in this study are sources of oxidative stress.

DETAILED DESCRIPTION:
The integrative vascular laboratory has recently observed that the small blood vessels in the skin (the cutaneous microvasculature) in obese (BMI>30kg/m2), but otherwise healthy individuals, require a greater amount of nitric oxide (NO) to achieve the same degree of dilation when compared to age, gender, and race matched lean (BMI<25kg/m2) individuals (34). In addition, it is well documented that African Americans have impaired blood vessel function which likely contributes to the elevated risk for developing a variety of cardiovascular and metabolic diseases including coronary artery disease, metabolic syndrome, hypertension and stroke in this population. The cutaneous circulation is recognized as a surrogate vascular bed for assessment of mechanisms underlying systemic vascular disease (7, 20, 22). This is particularly important as microvascular dysfunction is emerging as a critical step in the atherosclerotic process and a variety of conditions including hypertension, exercise intolerance, and insulin resistance (25). Furthermore, impaired cutaneous microvascular function mirrors impaired responses in other vascular beds (7, 12, 20, 22). A primary advantage to utilizing the cutaneous circulation is that it provides an accessible vascular bed through which processes of endothelial function can be systematically and mechanistically investigated, with virtually no risk, through thermal stimuli and local intra-dermal drug infusions. Mechanisms of impaired NO bioavailability have been assessed in various at-risk and diseased populations including, healthy aging, hypertension, postural tachycardia syndrome, hypercholesteremia, and chronic kidney disease (8, 16, 19, 24, 36, 37). Using approaches and techniques similar to those proposed in this application (see below) the findings have implicated that a number of factors, including elevated oxidative stress, contribute to the reduced bioavailability and/or action of NO (8, 16, 19, 24, 36, 37)

The recent findings suggest an impairment in the action of NO on the microvascular smooth muscle of obese young adults (34) as well as in college-aged otherwise healthy African Americans. Local heating is a common method to test nitric oxide-mediated vasodilation (3, 6, 31). Therefore, the investigators propose to test the following hypotheses:

1. Obesity results in impaired blood flow response to local heating and this will also be the case for African Americans.
2. Inhibition of superoxide, a common form of oxidative stress, augments the local heating response in obese individuals as well as in African Americans.
3. Inhibition of sources of superoxide, NADPH-oxidase and/or Xanthine-oxidase, augments skin blood flow local heating response in obese to that of their lean counterparts. This will also be the case for African Americans relative to their Caucasian American counterparts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (ages 18-35, both genders) will be recruited from the greater Arlington area to participate in the study.
* Must self-report both parents as either African American or Caucasian American.

Exclusion Criteria:

* Individuals who have donated more than 550 ml of blood within the past 8 weeks will not have blood drawn from them in this protocol. However, if they remain interested in the study, and otherwise meet the inclusion criteria, than we may still opt to proceed with data collection.
* Individuals with cardiovascular, neurological, and/or metabolic illnesses will be excluded from participating as well as individuals with a history of various diseases of the microvasculature including Reynaud's disease, cold-induced urticaria, cryoglobulinemia, etc.
* Subjects currently taking any prescription medications and individuals with a body mass index about 30 kg/m2) will be excluded.
* Pregnant subjects and children (i.e. younger than 18) will not be recruited for the study. Eligible females will be scheduled for days 2-7 of their menstrual cycle to account for hormonal effects on blood flow. A regular menstrual cycle is required to identify and schedule the study for the low hormone period, therefore females who lack a regular cycle will be excluded from the study. Females currently taking birth control are eligible, as long as they can be scheduled during a low-hormone "placebo" week. If their hormone do not contain a placebo week than these individuals will not be eligible for data collection. Females who are breast-feeding will also be eligible as there are no systemic or lasting effects of the proposed vasoactive agents.
* Given that smoking can affect the peripheral vasculature, current smokers and individuals who regularly smoked (>1 pack per two weeks) within the prior 2 years will be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Vasodilator Responses to Local Heating with Antioxidant Supplementation | Through study completion, an average of 1 year
  Assess the impact of oxidative stress on impaired vasodilation to local heating. This will be elicited using intradermal microdialysis infusions of apocynin, allopurinol, or tempol, all of which are vasoactive substances. The changes in skin blood flux will be quantified using laser Doppler fluxmetry. All changes in flux will be normalized and reported as a percentage of maximal flux.

CONTACTS AND LOCATIONS:
Locations (1):
- Engineering Research Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No